CLINICAL TRIAL: NCT05475678
Title: A Randomized, Open Label, Parallel Controlled, Multicenter Phase II Clinical Study of Carelizumab Combined With TCb (Docetaxel+Carboplatin) Versus TCb Neoadjuvant Therapy for Triple Negative Breast Cancer
Brief Title: Clinical Study of Camrelizumab Combined With TCb Versus TCb in Neoadjuvant Treatment of Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhenzhen Liu (Other Government)
Responsible Party: Sponsor-Investigator, Zhenzhen Liu, Director, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-011
Record Dates: First submitted 2022-07-19; First posted 2022-07-27 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; Camrelizumab
Keywords: Triple Negative Breast Cancer; Camrelizumab; Neoadjuvant chemotherapy; Pathological complete response rate; Disease-free survival
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — camrelizumab; Carboplatin; Docetaxel

STUDY DESIGN:
Intervention Model Description: The enrolled patients were randomly assigned to the experimental group and the control group in a ratio of 2:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- （Carrelizumab + TCb） regimen (Experimental): The experimental group received 6 cycles of TCb+carrelizumab (docetaxel 75mg/m2 on the first day + carboplatin AUC=6, on the first day; camrelizumab 200mg on the third day) regimen neoadjuvant chemotherapy, every 21 days is a cycle.
  Interventions: Drug: （Carrelizumab + TCb） regimen
- TCb regimen (Placebo Comparator): The control group received 6 cycles of TCb (docetaxel 75mg/m2 on the first day + carboplatin AUC=6 on the first day) regimen neoadjuvant chemotherapy, every 21 days as a cycle.
  Interventions: Drug: TCb regimen

INTERVENTIONS:
Drug: （Carrelizumab + TCb） regimen — Carrelizumab +docetaxel + carboplatin regimen
  Other Names: Carrelizumab +docetaxel + carboplatin
  Arms: （Carrelizumab + TCb） regimen
Drug: TCb regimen — docetaxel + carboplatin regimen
  Other Names: docetaxel + carboplatin
  Arms: TCb regimen

SUMMARY:
Triple-negative breast cancer (TNBC) is a special subtype of breast cancer that lacks the expression of ER, PR, and Her-2 proteins, accounting for 15%-20% of all breast cancers.TNBC patients do not benefit from endocrine therapy or HER-2-targeted therapy, but are sensitive to cytotoxic drug therapy.Although the survival of TNBC patients has improved significantly compared with the past, it is still the type with the worst prognosis among all subtypes of breast cancer. Methods and drugs to further improve the therapeutic effect of TNBC patients are still being explored.

Camrelizumab, a PD-1 inhibitor produced by Hengrui, has been approved for the treatment of various malignant tumors including advanced lung cancer, advanced liver cancer and advanced esophageal cancer. Shows good therapeutic effect and safety.

Therefore, this study intends to explore the superiority of camrelizumab on the basis of the less toxic anthracycline-free TCb regimen.In order to provide more effective and safe neoadjuvant therapy for lymph node-positive TNBC patients.

DETAILED DESCRIPTION:
This study mainly compared the efficacy and safety of 6*TCb (docetaxel+carboplatin)+carrelizumab regimen and 6*TCb regimen in neoadjuvant chemotherapy for triple-negative breast cancer.

Patients who met the inclusion criteria were randomly assigned to the experimental group and the control group in a 2:1 ratio.

* The experimental group received 6 cycles of TCb+carrelizumab (docetaxel 75mg/m2 on the first day + carboplatin AUC=6, on the first day; camrelizumab 200mg on the third day) regimen neoadjuvant chemotherapy, every 21 days is a cycle.
* The control group received 6 cycles of TCb (docetaxel 75mg/m2 on the first day + carboplatin AUC=6 on the first day) regimen neoadjuvant chemotherapy, every 21 days as a cycle.

The efficacy and safety of the two chemotherapy regimens on neoadjuvant chemotherapy for triple-negative breast cancer were evaluated by PCR, EFS, DFS, DDFS and ORR after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old
2. cT2 - cT4d, or cT1c with axillary lymph node metastasis confirmed clinically and pathologically；
3. Pathologically proven triple negative breast cancer:

   Triple-negative breast cancer is defined as:
   * Negative for ER and PR (IHC nuclear staining <10%)
   * Her-2 negative (IHC 0, 1+ without FISH, or IHC 2+ with no amplification by FISH)；
4. Has clinically measurable lesions:Measurable lesions on ultrasound, mammography, or MR (optional) within 1 month before randomization；
5. Organ and bone marrow function tests within 1 month before chemotherapy suggest no contraindications to chemotherapy；
6. Cardiac ultrasound EF value ≧55%；
7. Females of childbearing age, with a negative serum pregnancy test 14 days before randomization;
8. ECOG score≤1 point;
9. Sign informed consent；

Exclusion Criteria:

1. The patient has evidence of metastatic breast cancer；
2. For this disease, chemotherapy, endocrine therapy, targeted therapy, radiation therapy, etc. have been received;
3. The patient has a second primary malignancy other than adequately treated skin cancer;
4. The patient has been treated with anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death ligand 1 (anti-PD-L1) or anti-PD-L2 drugs, or other immunotherapy；
5. The patient has been diagnosed with immunodeficiency disease or autoimmune disease;
6. The patient has severe lung or heart disease;
7. The patient has active hepatitis B and C;
8. The patient has a history of organ transplantation or bone marrow transplantation;
9. pregnant or breastfeeding women;
10. The investigators considered chemotherapy contraindicated due to serious, uncontrolled other medical conditions.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR rate) | up to 24 weeks
  After neoadjuvant chemotherapy and surgery, the resected specimen (breast + axilla) was free of any invasive cancer (ie, ypT0/is, ypN0)

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | 5-10 years after surgery.
  EFS was defined as the time from randomization to any of the following events: disease progression during neoadjuvant therapy, local or distant recurrence, second primary malignancy (breast or other cancer), or death from any cause.
DFS | 5-10 years after surgery
  Disease-free Survival,From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause
Distant Disease Free Survival (DDFS) | 5-10 years after surgery
  DDFS is defined as the time from surgery to distant recurrence or death from any cause
Objective Response Rate (ORR) | Preoperative
  ORR is defined as the number of target lesion responders as assessed by MRI
number of adverse events | After each cycle of chemotherapy (21 days as 1 cycle)
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0

OTHER OUTCOMES:
Expression of PD-L1 | up to 24 weeks
  Differences in the benefits of carelizumab under different PD-L1 expression status
gene mutation rate | up to 24 weeks
  Predictive value of polygenic analysis in the population benefiting from camrelizumab

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Study Principal Investigator
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China